CLINICAL TRIAL: NCT01483417
Title: Multi-institution, Randomized Trial for Efficacy and Safety of Single Incision Laparoscopic Surgery (SILS) Versus Conventional Laparoscopic Hysterectomy for the Treatment of Uterine Myoma or Adenomyosis
Brief Title: Single Incision Laparoscopic Surgery (SILS) Versus Conventional Laparoscopic Hysterectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Joong Kim, Clinical Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-004
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2011-11

CONDITIONS: Uterine Myoma; Uterine Adenomyosis
Keywords: SILS; Laparoscopic hysterectomy; Cosmetic outcome; Pain
MeSH Terms: conditions — Myofibroma; Adenomyosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SILS (Experimental): Laparoscopic hysterectomy including LAVH, LH(a), and TLH using SILS port
  Interventions: Procedure: Single incision Laparoscopic hysterectomy
- Conventional multi-port laparoscopic hysterectomy (Active Comparator): 3-4 ports laparoscopic hysterectomy including LAVH, LH(a), or TLH
  Interventions: Procedure: Conventional laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Single incision Laparoscopic hysterectomy — SILS port
  Arms: SILS
Procedure: Conventional laparoscopic hysterectomy — 3-4 conventional ports
  Arms: Conventional multi-port laparoscopic hysterectomy

SUMMARY:
Multi-center prospective randomized trial of single port laparoscopic surgery (SILS) versus conventional 3-4 ports laparoscopic hysterectomy. Hypothesis is that conversion rate of SILS is not inferior to that of conventional approach.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic (dysmenorrhea, palpable mass, pelvic pain or discomfort urinary symptom, increasing size, menorrhagia) myomas or adenomyomas
* Uterine size < gestational age of 14 weeks
* Informed consent

Exclusion Criteria:

* Medical diseases such as heart failure, renal insufficiency, liver cirrhosis, pancreatitis, uncontrolled DM
* Huge uterine size > gestational age of 14 weeks

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | 1 week
  Conversion means that events required additional port(s) or open laparotomy

SECONDARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | 12 weeks
Postoperative pain | postop. 1 day, 1 week
  Measured by numeric rating score (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Heum Cho, MD, PhD, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (8):
- South Korea (8):
  - Keimyung University Dongsan Hospital, Deagu
  - Catholic Incheon Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Kangnam Cha Hospital, Seoul
  - Seoul Catholic Medical Center, Seoul
  - Yonsei University Medical Center, Seoul
  - Seoul University Bundang Hospital, Seungnam

REFERENCES:
- [Background] Kim TJ, Lee YY, Cha HH, Kim CJ, Choi CH, Lee JW, Bae DS, Lee JH, Kim BG. Single-port-access laparoscopic-assisted vaginal hysterectomy versus conventional laparoscopic-assisted vaginal hysterectomy: a comparison of perioperative outcomes. Surg Endosc. 2010 Sep;24(9):2248-52. doi: 10.1007/s00464-010-0944-y. Epub 2010 Feb 23. PMID 20177921
- [Background] Lee YY, Kim TJ, Kim CJ, Kang H, Choi CH, Lee JW, Kim BG, Lee JH, Bae DS. Single-port access laparoscopic-assisted vaginal hysterectomy: a novel method with a wound retractor and a glove. J Minim Invasive Gynecol. 2009 Jul-Aug;16(4):450-3. doi: 10.1016/j.jmig.2009.03.022. Epub 2009 May 31. PMID 19487164
- [Background] Jung YW, Lee M, Yim GW, Lee SH, Paek JH, Kwon HY, Nam EJ, Kim SW, Kim YT. A randomized prospective study of single-port and four-port approaches for hysterectomy in terms of postoperative pain. Surg Endosc. 2011 Aug;25(8):2462-9. doi: 10.1007/s00464-010-1567-z. Epub 2011 Feb 7. PMID 21298522
- [Background] Chen YJ, Wang PH, Ocampo EJ, Twu NF, Yen MS, Chao KC. Single-port compared with conventional laparoscopic-assisted vaginal hysterectomy: a randomized controlled trial. Obstet Gynecol. 2011 Apr;117(4):906-912. doi: 10.1097/AOG.0b013e31820c666a. PMID 21422864